CLINICAL TRIAL: NCT01991821
Title: Randomised, Double-blind, Placebo-controlled Phase III Study of APD421 (Amisulpride for IV Injection) as Prophylaxis Against Post-operative Nausea and Vomiting
Brief Title: European Phase III Study of APD421 in PONV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DP10014
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APD421 (Experimental): IV APD421 single dose
  Interventions: Drug: APD421
- Placebo (Placebo Comparator): IV placebo single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD421
  Arms: APD421
Drug: Placebo
  Arms: Placebo

SUMMARY:
A comparison of the efficacy of APD421 and placebo in the prevention of PONV in patients at moderate-to-high risk of PONV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients undergoing elective surgery (open or laparoscopic technique) under general anaesthesia, expected to last at least one hour from induction of anaesthesia to wound closure and expected to require at least one overnight stay in hospital

Exclusion Criteria:

* Patients scheduled for outpatient/day case surgery
* Patients scheduled to undergo intra-thoracic, transplant or central nervous system surgery
* Patients scheduled to receive only a local anaesthetic/regional neuraxial (intrathecal or epidural) block
* Patients who are expected to remain ventilated for a period after surgery
* Patients who are expected to need a naso- or orogastric tube in situ after surgery is completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Diemunsch, MD, Principal Investigator — Hôpital de Hautepierre
Locations (2):
- CHU de Hautepierre, Strasbourg, France
- University Hospitals of Würzburg, Würzburg, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 368 patients enrolled in the study, 21 patients were not randomised and not dosed. Of these, 3 withdrew their consent, 5 did not comply with the protocol procedures and 13 were not dosed for other unspecified reasons.
Groups:
- APD421: APD421 (amisulpride), at 5 mg given by single intravenous (IV) administration, by slow push over one to two minutes, at induction of anaesthesia.
- Placebo: Matching placebo, given by single IV administration, by slow push over one minute at the induction of anaesthesia.
Period: Overall Study
Arm/Group | APD421 | Placebo
Started | 169 | 178
Completed | 6 | 11
Not Completed | 163 | 167

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APD421 | Placebo | Total
Number analyzed (Participants) | 169 | 178 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (16.2) | 51.6 (14.9) | 51.6 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 154 | 301
  Male | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (no Emesis, Significant Nausea or Rescue Medication)
Description: The primary efficacy analysis was a comparison of the incidence of Complete Response (absence of PONV1) in the 0-24-hour period after surgery, between the active treatment group and the placebo group using Pearson square test with Yates's continuity correction at a two-sided significance level of 5%.
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 95 | 83
Statistical Analysis 1: Comparison: APD421 vs Placebo; The primary efficacy analysis was a complete response which is defined as protection from PONV1, which was absence of any episode of emesis, significant nausea or use of rescue medication with the first 24 hours post-operatively; Test type: Superiority; p = 0.093, Chi-squared, Corrected — The complete response of the primary efficacy analysis occurred in 95 patients (56.2%; 95% confidence interval [CI] 48.4 - 63.8%) in the APD421 group and 83 patients (46.6%; 95% CI 39.1- 54.2%) in the placebo group; Pearson square test with Yates's continuity correction and with the two- sided significance level of 5%

2. Secondary Outcome: Complete Response (no Emesis or Rescue Medication)
Time Frame: 24 hrs after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 100 | 89
Statistical Analysis 1: Comparison: APD421 vs Placebo; Test type: Superiority; p = 0.059, Chi-squared, Corrected — Two-sided, significance threshold = 0.05

3. Secondary Outcome: Total Response (no Emesis, Nausea or Rescue Medication)
Time Frame: 24 hrs after end of surgery
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 87 | 73
Statistical Analysis 1: Comparison: APD421 vs Placebo; Test type: Superiority; p = 0.053, Chi-squared, Corrected — Two-sided, significance threshold = 0.05

4. Secondary Outcome: Incidence of Emesis (Vomiting/Retching)
Description: An assessment of a participant experiencing an episode of emesis (vomiting/ retching) or received anti-emetic rescue medication during the 24hours after the completion of the surgery
Time Frame: 24 hours after end of surgeryry
Measure: Count of Participants; unit: Participants
Groups:
- APD421 at 5mg: IV 5mg APD421 single dose
- Placebo: IV placebo single dose
  Placebo
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 34 | 46
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.26, Chi-squared, Corrected — Two-sided, significance threshold = 0.05

5. Secondary Outcome: Incidence of Nausea
Description: Count of patients experiencing an episode of nausea scored ≥ 1 of 0-10 verbal response scale during the 24 hours period after the completion of surgery
Time Frame: 24 hours after end of surgery
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 at 5mg | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 75 | 98
Statistical Analysis 1: Comparison: APD421 at 5mg vs Placebo; Test type: Superiority; p = 0.06, Chi-squared, Corrected — Two-sided, significance threshold = 0.05

6. Secondary Outcome: Incidence of Significant Nausea
Description: Count of participants with nausea score ≥ 4 on 0-10 verbal response scale
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 63 | 84
Statistical Analysis 1: Comparison: APD421 vs Placebo; Test type: Superiority; p = 0.079, Chi-squared, Corrected — Two-sided, significance threshold = 0.05

7. Secondary Outcome: Use of Rescue Medication
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 | Placebo
Number analyzed (Participants) | 169 | 178
Participants | 62 | 82
Statistical Analysis 1: Comparison: APD421 vs Placebo; Test type: Superiority; p = 0.096, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Any AE that is serious occurring during the course of the study, irrespective of the treatment received by the subject must be reported to the pharmacovigilance provider within 24hours of it's recognition
Groups:
- APD421 at 5mg: APD421 at 5mg given by single intravenous (IV) administration, by slow push over one to two minutes at induction of anaesthesia.
- Placebo: APD421 Placebo given by single IV administration by slow push over one minute at induction of anaesthesia.
Arm/Group | APD421 at 5mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/178
Serious Adverse Events (participants affected / at risk) | 3/169 | 4/178
Other Adverse Events (participants affected / at risk) | 91/169 | 178/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 at 5mg (N=169) | Placebo (N=178)
Anastomic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 at 5mg (N=169) | Placebo (N=178)
Procedural Pain (Injury, poisoning and procedural complications) | 91 (91) | 92 (92)
Constipation (Gastrointestinal disorders) | 16 (16) | 9 (9)
Flatulence (Gastrointestinal disorders) | 18 (18) | 16 (16)
Nausea (Gastrointestinal disorders) | 20 (20) | 18 (18)
Blood Prolactin Increased (Investigations) | 18 (18) | 2 (2)
Hypotension (Vascular disorders) | 9 (9) | 14 (14)
Headache (Nervous system disorders) | 14 (14) | 9 (9)
Sleep Disorder (Psychiatric disorders) | 7 (7) | 9 (9)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 9 (9)

LIMITATIONS AND CAVEATS:
There are no limitations and caveats with this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days